CLINICAL TRIAL: NCT01261949
Title: Effectiveness of Low Frequency Combined Frontal and Temporal Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Chronic Tinnitus
Brief Title: Combined Low Frequency Frontal and Temporal rTMS Treatment in Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, Ph.D., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uni-Reg-rTMS-Tinnitus-02
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Tinnitus
Keywords: Tinnitus; chronic subjective tinnitus; transcranial magnetic stimulation; sensation disorders; hearing disorders
MeSH Terms: conditions — Tinnitus; Sensation Disorders; Hearing Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined frontal and temporal rTMS (Experimental): Combined low frequency frontal and temporal transcranial magnetic stimulation of auditory cortex and right DLPFC
  Interventions: Device: Combined frontal and temporal rTMS
- Temporal low frequency rTMS (Experimental): temporal low frequency rTMS of auditory cortex
  Interventions: Device: Temporal low frequency rTMS

INTERVENTIONS:
Device: Combined frontal and temporal rTMS — Experimental repetitive transcranial magnetic stimulation (Alpine Biomed Mag Pro Option): 1000 stimuli of 1Hz rTMS over the right DLPFC (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over the left temporal cortex DLPFC (110% motor threshold)
  Arms: Combined frontal and temporal rTMS
Device: Temporal low frequency rTMS — Experimental repetitive transcranial magnetic stimulation (Alpine Biomed Mag Pro Option): 2000 stimuli of 1 Hz rTMS over the left temporal cortex (110% motor threshold)
  Arms: Temporal low frequency rTMS

SUMMARY:
Transcranial Magnetic Stimulation is used to modulate the auditory neural pathways caused by hearing loss and leading to the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Treatment is difficult. Most available therapies focus on habituation rather than treating the cause. Tinnitus is thought to be generated in the brain, as a result of functional reorganization of auditory neural pathways and tonotopic maps in the central auditory system, following damage to the peripheral auditory system. Low-frequency rTMS has been investigated for the treatment of hyperexcitability disorders such as auditory hallucinations and tinnitus. Pilot data indicate that the beneficial effect of low-frequency rTMS can be enhanced by low frequency rTMS of the right dorsolateral prefrontal cortex (DLPFC). In the proposed study we investigate whether low frequency rTMS of the DLPFC improves therapeutic efficacy of low-frequency rTMS on tinnitus in a controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subjective chronic tinnitus
* Duration of tinnitus more than 3 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery;
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Prior treatment with TMS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Questionnaire of Goebel and Hiller | Baseline, Day 12

SECONDARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller, Tinnitus Handicap Inventory (THI), Tinnitus Severity Scale and TBF-12 | Baseline vs. all follow-up visits
Change of depressive symptoms as measured by the Beck Depression Inventory (BDI) | Baseline vs. all follow-up visits
Change in quality of life as measured by the WHOQoL | Baseline vs. all follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Principal Investigator — University of Regensburg - Dep. of Psychiatry
Locations (1):
- University of Regensburg - Dept of Psychiatry, Regensburg, Bavaria, Germany

REFERENCES:
- [Result] Kreuzer PM, Landgrebe M, Schecklmann M, Poeppl TB, Vielsmeier V, Hajak G, Kleinjung T, Langguth B. Can Temporal Repetitive Transcranial Magnetic Stimulation be Enhanced by Targeting Affective Components of Tinnitus with Frontal rTMS? A Randomized Controlled Pilot Trial. Front Syst Neurosci. 2011 Nov 4;5:88. doi: 10.3389/fnsys.2011.00088. eCollection 2011. PMID 22069382
- See also: Tinnitus Research and Treatment Center at the University of Regensburg — http://www.tinnituszentrum-regensburg.de